CLINICAL TRIAL: NCT01010581
Title: A Randomized, Double Blind, Placebo-Controlled, Phase II Study to Evaluate Efficacy, Safety, and Pharmacokinetics of SC12267 (35 mg) in Combination With Methotrexate Compared to Methotrexate Alone in Patients With Rheumatoid Arthritis
Brief Title: SC12267 (4SC-101) in Combination With Methotrexate in Patients With Rheumatoid Arthritis
Acronym: COMPONENT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: 4SC AG (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SC12267-5-2009
Record Dates: First submitted 2009-11-09; First posted 2009-11-10 (Estimated); Last update posted 2012-03-01 (Estimated); Status verified 2012-02

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; SC12267; 4SC-101; Methotrexate; Phase II
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — vidofludimus; Methotrexate; Folic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- SC12267 (4SC-101) + Methotrexate (Experimental)
  Interventions: Drug: SC12267 (4SC-101); Drug: Methotrexate; Drug: Folic Acid
- Placebo + Methotrexate (Placebo Comparator)
  Interventions: Drug: Placebo; Drug: Methotrexate; Drug: Folic Acid

INTERVENTIONS:
Drug: SC12267 (4SC-101) — oral administration
  Arms: SC12267 (4SC-101) + Methotrexate
Drug: Placebo — oral administration
  Arms: Placebo + Methotrexate
Drug: Methotrexate — oral administration
Drug: Folic Acid — oral administration

SUMMARY:
The purpose of the study is to determine the efficacy, safety and pharmacokinetics of SC12267 (4SC-101, 35 mg) in combination with methotrexate in comparison to methotrexate alone in the treatment of patients suffering from Rheumatoid Arthritis.

ELIGIBILITY:
Main Inclusion Criteria:

* Patients with active RA of functional classes I, II or III according to the criteria of American Rheumatism Association for RA
* DAS28(ESR) ≥ 4.5 (DAS28 formula with 4 variables using ESR)
* Patients who have received weekly doses of MTX (10-25 mg/week) for a minimum of 3 months prior to Day 1 dosing, and who have received a stable MTX dose of 10-25 mg/week without any change in route or change in folic acid supplementation for at least 6 weeks prior to Day 1 dosing
* Patients may receive up to 10 mg/day of oral prednisolone or steroid equivalent. Dose must have been stable for at least 30 days and must not be changed during the washout, screening and treatment periods, unless dictated by tolerability requirements

Main Exclusion Criteria:

* Patients with RA of functional classes IV according to the criteria of American Rheumatism Association for RA
* Patients who have received any of the following treatments must abide by the indicated washout period:

  1. Leflunomide requires a 6 month washout period prior to Day 1 dosing
  2. Oral or injectable gold, azathioprine, penicillamine, anakinra require a 30 day washout period prior to Day 1 dosing
  3. Cyclosporine, abatacept, etanercept, adalimumab, infliximab, and rituximab require a 60 day washout period prior to Day 1 dosing
  4. Cyclophosphamide requires a 180 day washout period prior to Day 1 dosing
  5. Parenteral or intra-articular corticosteroids require a 30 day washout period prior to Day 1 dosing
* Receipt of the following drugs within 4 weeks prior to dosing:

  1. Sulfasalazine
  2. Hydroxychloroquine
  3. Use of corticosteroids > 10 mg/day

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 266 (Actual)
Dates: Start 2009-11; Primary Completion 2011-04 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Efficacy of SC12267 (4SC-101) in combination with methotrexate in patients with RA | 13 weeks

SECONDARY OUTCOMES:
Evaluation of the safety of the combination of SC12267 (4SC-101) and methotrexate in patients with RA | 13 weeks
Evaluation of the plasma concentration (trough value) of SC12267 (4SC-101) after once daily application in combination with methotrexate after once weekly administration. | 13 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Stanisław Sierakowski, Prof. MD, Principal Investigator — Centrum Miriada, Prywatny Gabinet Specjalistyczny, Bialystok, Poland
Locations (27):
- Bulgaria (5):
  - MHAT "Kaspela" Department of Rheumatology, Plovdiv
  - Diagnostic Consulting Centre "Sv. Anna", Sofia
  - Military Medical Academy, Sofia
  - National Multiprofile Transport Hospital "Tsar Boris III" Internal Clinic, Sofia
  - UMHAT "Sveti Ivan Rilski", Sofia
- Czechia (3):
  - Rheumatology Outpatient Clinic, Hlučín
  - Diagnostic Center Mediscan, Prague
  - Institute of Rheumatology, Prague
- Poland (12):
  - Centrum Miriada, Prywatny Gabinet Specjalistyczny, Bialystok
  - Mazowieckie Centrum Badań Klinicznych s.c., Grodzisk Mazowiecki
  - Śląskie Centrum Osteoporozy, Katowice
  - Specjalistyczny Ośrodek ALL-MED, Krakow
  - NZOZ Reumed, Lublin
  - Prof. Dr Hab. n. m. Leszek Szczepański, Lublin
  - Poznański Ośrodek Medyczny NOVAMED, Poznan
  - Wojewódzki Szpital Reumatologiczny, Sopot
  - NZOZ "Nasz Lekarz", Torun
  - Centrum Leczenia Chorób Cywilizacyjnych Sp. z o. o. S. K. A., Warsaw
  - Centrum Medyczne Osteomed NZOZ Lecznica Specjalistów, Warsaw
  - NZOZ Materia Medica, Wroclaw
- Romania (7):
  - Clinic Hospital Sf. Maria, Bucharest
  - Emergency Hospital "Prof. Dr. Gerota", Bucharest
  - SC Duomedical, Bucharest
  - SC Ianuli Med Consult, Bucharest
  - County Hospital Cluj - Rheumatology clinic, Cluj-Napoca
  - Clinical County Hospital of Targoviste, Targoviste, Dambovita
  - Private Practice Prof. Dr. Mioara Banciu, Timișoara

REFERENCES:
- [Derived] Muehler A, Kohlhof H, Groeppel M, Vitt D. The Selective Oral Immunomodulator Vidofludimus in Patients with Active Rheumatoid Arthritis: Safety Results from the COMPONENT Study. Drugs R D. 2019 Dec;19(4):351-366. doi: 10.1007/s40268-019-00286-z. PMID 31621054
- [Derived] Kulkarni OP, Sayyed SG, Kantner C, Ryu M, Schnurr M, Sardy M, Leban J, Jankowsky R, Ammendola A, Doblhofer R, Anders HJ. 4SC-101, a novel small molecule dihydroorotate dehydrogenase inhibitor, suppresses systemic lupus erythematosus in MRL-(Fas)lpr mice. Am J Pathol. 2010 Jun;176(6):2840-7. doi: 10.2353/ajpath.2010.091227. Epub 2010 Apr 22. PMID 20413687